CLINICAL TRIAL: NCT04151966
Title: Evaluation of Potential Myocardial Injury Following Elective Direct Current Cardioversion for Atrial Arrhythmias
Brief Title: Myocardial Injury Following Elective Direct Current Cardioversion for Atrial Arrhythmias
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Allan S. Jaffe, Principal Investigator, Mayo Clinic
Other Study IDs: 19-004287
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Cardioversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum or plasma samples remaining after initial analysis will be frozen and stored at -80 degrees Celsius for 120 months (10 years). These samples may be used if there are new and more sensitive biomarkers of myocardial injury that become available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardioversion Group: Subjects scheduled to undergo direct current cardioversion (DCCV) as part of the clinical plan of care
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Blood sample collection for markers of myocardial injury

SUMMARY:
Researchers are trying to determine if heart injury occurs in subjects who undergo direct current cardioversion.

DETAILED DESCRIPTION:
External transthoracic direct current (DC) cardioversion is a commonly used method of terminating cardiac arrhythmias. Conventional wisdom indicates that external DC cardioversion causes myocardial injury. Previous research has shown that DC cardioversion resulted in myocardial injury as evidenced by increased levels of cardiac troponin, even though those changes were modest. Many of these studies evaluated monophasic defibrillators and older, less sensitive cardiac troponin assays. The current standard is now to use modern biphasic defibrillators and new high sensitivity cardiac troponin assays (hs-cTnT). It is conceivable that the newer defibrillators may not cause myocardial injury. It would be important to understand if myocardial injury occurs in this setting and its approximate magnitude as it would the interpretation of hs-cTnT values in patients and therefore influenced diagnoses. It may be if a threshold energy level can be identified that is would also influence the choice of energy used to deliver the shock in this situation.

A previous preliminary study documented no evidence of myocardial injury after elective DC cardioversion with modern day defibrillators. We aim to validate and expand that study here at Mayo Clinic Rochester.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing elective direct current cardioversion, either externally or via the patient's internal cardioverter-defibrillator

Exclusion Criteria:

* Patients under age 18
* Patients with myocardial infarction, coronary artery bypass grafting or any invasive cardiac procedure in the previous six weeks
* Pregnant patients
* Patients who cannot provide informed consent because of cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and females age 18 and above identified from the electronic medical record (EMR) calendar of patients scheduled for an elective direct current cardioversion.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Myocardial injury | Baseline, 6-24 hours post procedure
  Changes in high sensitivity cardiac troponin T (hs-cTnT) or troponin I (hs-cTnI) assay

CONTACTS AND LOCATIONS:
Overall Officials: Allan S Jaffe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials